CLINICAL TRIAL: NCT03690869
Title: A Safety and Pharmacokinetic Study of Single Agent REGN2810 in Pediatric Patients With Relapsed or Refractory Solid or Central Nervous System (CNS) Tumors and a Safety and Efficacy Trial of REGN2810 in Combination With Radiotherapy in Pediatric Patients With Newly Diagnosed Diffuse Intrinsic Pontine Glioma, Newly Diagnosed High-Grade Glioma, or Recurrent High-Grade Glioma
Brief Title: REGN2810 in Pediatric Patients With Relapsed, Refractory Solid, or Central Nervous System (CNS) Tumors and Safety and Efficacy of REGN2810 in Combination With Radiotherapy in Pediatric Patients With Newly Diagnosed or Recurrent Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Pacific Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1690; PNOC 013 (CC#160825) (Other: Pacific Pediatric Neuro-Oncology Consortium (PNOC))
Record Dates: First submitted 2018-09-17; First posted 2018-10-01 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Relapsed Solid Tumor; Refractory Solid Tumor; Relapsed Central Nervous System Tumor; Refractory Central Nervous System Tumor; Diffuse Intrinsic Pontine Glioma; High Grade Glioma
Keywords: Newly Diagnosed; Recurrent; Refractory
MeSH Terms: conditions — Central Nervous System Neoplasms; Diffuse Intrinsic Pontine Glioma; Glioma; Recurrence | interventions — cemiplimab; Maintenance; Congresses as Topic; Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 (Experimental): Patients in both the Solid Tumor Cohort and the CNS Cohort will receive cemiplimab monotherapy. Each Cohort will have 2 subgroups by age (0 to <12 years, 12 to <18 years).
  Interventions: Drug: cemiplimab (monotherapy)
- Efficacy with Newly Diagnosed DIPG (Experimental): ≥ 3 to < 12 years cohort and 12 to ≤ 25 years cohort with combination of cemiplimab and radiation therapy
  Interventions: Drug: cemiplimab (maintenance); Radiation: Conventional or hypofractionated
- Efficacy with Newly Diagnosed HGG (Experimental): ≥ 3 to < 12 years cohort and 12 to ≤ 25 years cohort with combination of cemiplimab and radiation therapy
  Interventions: Drug: cemiplimab (maintenance); Radiation: Conventional or hypofractionated
- Efficacy with Recurrent HGG (Experimental): ≥ 3 to < 12 years cohort and 12 to ≤ 25 years cohort with combination of cemiplimab and radiation therapy
  Interventions: Drug: cemiplimab (maintenance); Radiation: Re-irradiation

INTERVENTIONS:
Drug: cemiplimab (monotherapy) — To be administered intravenously as monotherapy in Phase 1
  Other Names: REGN2810; Libtayo
  Arms: Phase 1
Drug: cemiplimab (maintenance) — To be administered intravenously in combination with radiation and then used as maintenance therapy
  Other Names: REGN2810; Libtayo
  Arms: Efficacy with Newly Diagnosed DIPG; Efficacy with Newly Diagnosed HGG; Efficacy with Recurrent HGG
Radiation: Conventional or hypofractionated — Combined with cemiplimab IV administration
  Arms: Efficacy with Newly Diagnosed DIPG; Efficacy with Newly Diagnosed HGG
Radiation: Re-irradiation — Combined with cemiplimab IV administration
  Arms: Efficacy with Recurrent HGG

SUMMARY:
Phase 1:

* To confirm the safety and anticipated recommended phase 2 dose (RP2D) of REGN2810 (cemiplimab) for children with recurrent or refractory solid or Central Nervous System (CNS) tumors
* To characterize the pharmacokinetics (PK) of REGN2810 given in children with recurrent or refractory solid or CNS tumors

Phase 2 (Efficacy Phase):

* To confirm the safety and anticipated RP2D of REGN2810 to be given concomitantly with conventionally fractionated or hypofractionated radiation among patients with newly diagnosed diffuse intrinsic pontine glioma (DIPG)
* To confirm the safety and anticipated RP2D of REGN2810 given concomitantly with conventionally fractionated or hypofractionated radiation among patients with newly diagnosed high-grade glioma (HGG)
* To confirm the safety and anticipated RP2D of REGN2810 given concomitantly with re-irradiation in patients with recurrent HGG
* To assess PK of REGN2810 in pediatric patients with newly diagnosed DIPG, newly diagnosed HGG, or recurrent HGG when given in combination with radiation
* To assess anti-tumor activity of REGN2810 in combination with radiation in improving overall survival at 12 months (OS12) among patients with newly diagnosed DIPG
* To assess anti-tumor activity of REGN2810 in combination with radiation in improving progression-free survival at 12 months (PFS12) among patients with newly diagnosed HGG
* To assess anti-tumor activity of REGN2810 in combination with radiation in improving overall survival at OS12 among patients with recurrent HGG

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 0 to <18 years of age (Phase 1)
2. Age ≥3 and ≤25 years of age (Efficacy Phase)
3. Karnofsky performance status ≥50 (patients >16 years) or Lansky performance status ≥50 (patients ≤ 16 years)
4. Life expectancy >8 weeks
5. Adequate Bone Marrow Function
6. Adequate Renal Function
7. Adequate Liver Function
8. Adequate Neurologic Function

Key Exclusion Criteria:

1. Patients with bulky metastatic disease of the CNS causing Uncal herniation or symptomatic midline shift, significant, symptomatic mass effect, or uncontrolled neurological symptoms such as seizures or altered mental status
2. Patients with metastatic spine disease and gliomatosis as documented by diffuse involvement of >2 lobes
3. Patients who are receiving any other investigational anticancer agent(s)
4. Patients on greater than dexamethasone 0.1 mg/kg/day (maximum 4 mg/day) or equivalent dose in alternate corticosteroid, or actively undergoing corticosteroid dose escalation in the last 7 days
5. Patients with a history of allogeneic stem cell transplant
6. Prior treatment with an agent that blocks the PD-1/PD-L1/PD-L2 pathway

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (20):
- United States (20):
  - Children's Hospital Los Angeles (CHLA), Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's National Health System (Children's National Medical Center), Washington D.C., District of Columbia
  - University of Florida- Neurosurgery, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins - Pediatric Oncology, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute/ Boston Children's Hospital, Boston, Massachusetts
  - C. S. Mott/University of Michigan, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota / Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University (OHSU) - Doernbecher Children's Hospital, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer & Hematology Centers Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 65 participants were screened; 57 participants were enrolled and had received at least 1 dose of REGN2810 at time of study termination (Sponsor decision)
Groups:
- SOLID TUMOR < 12 yr REGN2810 3mg/kg: Phase 1 (Cohort A) SOLID TUMOR < 12 yr REGN2810 3 milligrams/kilogram (mg/kg) every two weeks (Q2W)
- SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg: Phase 1 (Cohort B) SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg (Q2W)
- CNS TUMOR <12 yr REGN2810 3mg/kg: Phase 1 (Cohort C1) Central Nervous System (CNS) TUMOR <12 yr REGN2810 3mg/kg (Q2W)
- CNS TUMOR <12 yr REGN2810 4.5mg/kg: Phase 1 (Cohort C2) CNS TUMOR <12 yr REGN2810 4.5mg/kg (Q2W)
- CNS TUMOR 12 to <18 yr REGN2810 3mg/kg: Phase 1 (Cohort D) CNS TUMOR 12 to <18 yr REGN2810 3mg/kg (Q2W)
- ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy: Efficacy Phase (Cohort E) ndDIPG <12 yr REGN2810 4.5mg/kg (Q2W) + Radiotherapy (pre-specified to be assessed regardless of which radiation therapy)
- ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy: Efficacy Phase (Cohort F) ndDIPG >=12 yr REGN2810 3mg/kg (Q2W) + Radiotherapy (pre-specified to be assessed regardless of which radiation therapy)
- ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy: Efficacy Phase (Cohort H) ndHGG >=12 yr REGN2810 3mg/kg (Q2W) + Radiotherapy (pre-specified to be assessed regardless of which radiation therapy)
- rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation: Efficacy Phase (Cohort I) rHGG <12 yr REGN2810 4.5mg/kg (Q2W) + Re-Irradiation
- rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation: Efficacy Phase (Cohort J) rHGG >= 12 yr REGN2810 3mg/kg (Q2W) + Re-Irradiation
Period: Overall Study
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Started | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 11 | 1 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Death | 1 | 1 | 1 | 4 | 2 | 5 | 3 | 2 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Treatment | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 7 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Subject Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CNS TUMOR <12 yr REGN2810 3mg/kg: Phase 1 (Cohort C1) CNS TUMOR <12 yr REGN2810 3mg/kg (Q2W)
- Total: Total of all reporting groups
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation | Total
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (5.29) | 13.4 (1.95) | 7.7 (1.53) | 7.1 (2.26) | 15.0 (1.00) | 4.8 (1.83) | 15.4 (2.41) | 16.4 (3.63) | 8.0 (0) | 16.3 (3.01) | 12.1 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4 | 2 | 4 | 4 | 4 | 1 | 2 | 25
  Male | 2 | 3 | 2 | 5 | 3 | 2 | 1 | 8 | 0 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 2 | 3 | 3 | 1 | 5 | 1 | 3 | 21
  Not Hispanic or Latino | 3 | 2 | 3 | 7 | 2 | 1 | 4 | 6 | 0 | 5 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 3 | 3 | 3 | 5 | 3 | 2 | 4 | 12 | 1 | 4 | 40
    Black or African American | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 6
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Unknown | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 4
    Not reported | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are AEs that developed or worsened during the on-treatment period and any treatment-related AEs that occur during the post-treatment period but prior to initiation of other anticancer therapy. Number of TEAEs reported.
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Population: Safety analysis set (SAF): All enrolled participants who have received any study treatment (at least one dose of any component of study treatment in a combination therapy) in each study phase. Participants analyzed according to the study treatment received (as treated).
Measure: Number; unit: Events
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Events | 19 | 42 | 24 | 56 | 49 | 108 | 102 | 222 | 28 | 175

2. Primary Outcome: Number of Severe (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] Grade 3/4/5) TEAEs
Description: NCI CTCAE version 4.0 was utilized for AE grading of severity: Grade 1 (Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 (Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 (Life-threatening consequences; urgent intervention indicated); Grade 5 (Death related to AE). Number of NCI grade 3/4/5 Treatment-Emergent Adverse Events (AEs) reported
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Events | 3 | 5 | 0 | 9 | 4 | 25 | 8 | 19 | 4 | 16

3. Primary Outcome: Number of Treatment-emergent Sponsor Identified Immune-related Adverse Events (irAEs)
Description: Number of sponsor-identified irAEs (all grades) reported.
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Events | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 9 | 0 | 9

4. Primary Outcome: Number of Severe (NCI CTCAE Grade 3/4/5) Treatment-emergent Sponsor Identified irAEs
Description: Number of severe treatment-emergent sponsor-identified irAEs reported.
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Events | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1

5. Primary Outcome: Number of Treatment-emergent AEs of Special Interest (AESI)
Description: AEs of special interest (AESI) are AEs required to be monitored, documented, and managed in a pre-specified manner as described in the protocol. Number of treatment-emergent AESI reported.
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Events | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 4 | 0 | 8

6. Primary Outcome: Number of NCI Grade 3/4/5 Treatment-emergent AESI
Description: Number of NCI grade 3/4/5 treatment-emergent AESI reported
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Events | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 4 | 0 | 6

7. Primary Outcome: Number of Participants With Any TEAE Resulting in Death
Description: Number of participants with any TEAE resulting in death reported
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With at Least One Lab Abnormality (NCI-CTCAE All Grades) in Hematology, Electrolytes, Liver, Chemistry
Description: Number of participants with new or worsened laboratory abnormalities (NCI-CTCAE All Grades) reported in Hematology, Electrolytes, Liver, Chemistry; Grade 1 (Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 (Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 (Life-threatening consequences; urgent intervention indicated); Grade 5 (Death related to AE).
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Participants
  ≥ 1 lab abnormality (All Grades) Hematology | 3 | 4 | 3 | 7 | 3 | 6 | 4 | 11 | 1 | 8
  ≥ 1 lab abnormality (All Grades) Electrolytes | 3 | 3 | 0 | 5 | 2 | 6 | 4 | 9 | 1 | 7
  ≥ 1 lab abnormality (All Grades) Liver | 1 | 2 | 0 | 5 | 3 | 4 | 5 | 7 | 1 | 5
  ≥ 1 lab abnormality (All Grades) Chemistry | 3 | 5 | 3 | 6 | 4 | 6 | 4 | 10 | 1 | 7

9. Primary Outcome: Number of Participants Who Developed Dose Limiting Toxicities (DLTs) (Phase 1)
Description: Number of participants who developed dose limiting toxicities (DLTs) in phase 1 reported
Time Frame: Baseline to 28 days
Population: Only Phase 1 participants that were eligible for Dose Limiting Toxicity evaluation.
Measure: Number; unit: Participants
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg
Number analyzed (Participants) | 2 | 5 | 3 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants Who Developed DLTs (Efficacy Phase)
Time Frame: Up to 4 weeks post radiation therapy
Population: Only Efficacy Phase participants that were eligible for Dose Limiting Toxicity evaluation.
Measure: Number; unit: Participants
Groups:
- Cohort E Efficacy Phase ndDIPG (DLT AS): Participants (3 to <12 years) with ndDIPG; DLT analysis set
- Cohort F Efficacy Phase ndDIPG (DLT AS): Participants (12 to 25 years) with ndDIPG; DLT analysis set
- Cohort H Efficacy Phase ndHGG (DLT AS): Participants (12 to 25 years) with ndHGG; DLT analysis set
- Cohort I Efficacy Phase rHGG (DLT AS): Participants (3 to <12 years) with rHGG; DLT analysis set
- Cohort J Efficacy Phase rHGG (DLT AS): Participants (12 to 25 years) with rHGG; DLT analysis set
Arm/Group | Cohort E Efficacy Phase ndDIPG (DLT AS) | Cohort F Efficacy Phase ndDIPG (DLT AS) | Cohort H Efficacy Phase ndHGG (DLT AS) | Cohort I Efficacy Phase rHGG (DLT AS) | Cohort J Efficacy Phase rHGG (DLT AS)
Number analyzed (Participants) | 6 | 5 | 6 | 1 | 6
Participants | 1 | 1 | 0 | 0 | 1

11. Primary Outcome: Elimination Half-life (t1/2) of Functional Cemiplimab (REGN2810) in Serum
Time Frame: Up to 24 months
Population: Cohorts used for pharmacokinetic endpoints were based on age and/or tumor type. Radiation type was collected, but not used for assessment; Due to sparse sampling, elimination half-life could not be calculated.
Measure: Median (Full Range); unit: milligrams/Liter (mg/L)
Groups:
- Cohort A Phase 1 ST 3mg/kg Q2W (PKAS): Participants (0 to <12 years) with recurrent or refractory ST received REGN2810 3mg/kg Q2W; Pharmacokinetic Analysis Set (PKAS)
- Cohort B Phase 1 ST 3mg/kg Q2W (PKAS): Participants (12 to <18 years) with recurrent or refractory ST received REGN2810 3mg/kg Q2W; PKAS
- Cohort C Phase 1 CNS 3mg/kg Q2W (PKAS): Participants (0 to <12 years) with recurrent or refractory CNS tumors received REGN2810 3mg/kg Q2W; PKAS
- Cohort C Phase 1 CNS 4.5mg/kg Q2W (PKAS): Participants (0 to <12 years) with recurrent or refractory CNS tumors received REGN2810 4.5mg/kg Q2W; PKAS
- Cohort D Phase 1 CNS 3mg/kg Q2W (PKAS): Participants (12 to <18 years) with recurrent or refractory CNS received REGN2810 3mg/kg Q2W; PKAS
- Cohort E Efficacy Phase ndDIPG 4.5mg/kg Q2W (PKAS): Participants (3 to <12 years) with ndDIPG received REGN2810 4.5mg/kg Q2W; PKAS
- Cohort F Efficacy Phase ndDIPG 3mg/kg Q2W (PKAS): Participants (12 to 25 years) with ndDIPG received REGN2810 3mg/kg Q2W; PKAS
- Cohort H Efficacy Phase ndHGG 3mg/kg Q2W (PKAS): Participants (12 to 25 years) with ndHGG received REGN2810 3mg/kg Q2W; PKAS
- Cohort I Efficacy Phase rHGG 4.5mg/kg Q2W (PKAS): Participants (3 to <12 years) with rHGG received REGN2810 4.5mg/kg Q2W; PKAS
- Cohort J Efficacy Phase rHGG 3mg/kg Q2W (PKAS): Participants (12 to 25 years) with rHGG received REGN2810 3mg/kg Q2W; PKAS
Arm/Group | Cohort A Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort B Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 4.5mg/kg Q2W (PKAS) | Cohort D Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort E Efficacy Phase ndDIPG 4.5mg/kg Q2W (PKAS) | Cohort F Efficacy Phase ndDIPG 3mg/kg Q2W (PKAS) | Cohort H Efficacy Phase ndHGG 3mg/kg Q2W (PKAS) | Cohort I Efficacy Phase rHGG 4.5mg/kg Q2W (PKAS) | Cohort J Efficacy Phase rHGG 3mg/kg Q2W (PKAS)
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 4 | 12 | 1 | 7
milligrams/Liter (mg/L) | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated. | NA [NA to NA] — Due to sparse sampling, elimination half-life could not be calculated.

12. Primary Outcome: Trough Concentration (Ctrough) of Functional Cemiplimab (REGN2810) in Serum
Description: Ctrough (trough concentration) of functional cemiplimab in serum reported.
Time Frame: Up to Week 16
Population: Pharmacokinetic Analysis Set (PKAS): All treated participants who received any amount of study drug (SAF) and had at least 1 non-missing functional cemiplimab measurement following the first dose of cemiplimab (based on actual treatment received [as treated]); Cohorts used for pharmacokinetic endpoints were based on age and/or tumor type.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Cohort A Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort B Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort D Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 4.5mg/kg Q2W (PKAS) | Cohort F Efficacy Phase ndDIPG 3mg/kg Q2W (PKAS) | Cohort H Efficacy Phase ndHGG 3mg/kg Q2W (PKAS) | Cohort J Efficacy Phase rHGG 3mg/kg Q2W (PKAS) | Cohort E Efficacy Phase ndDIPG 4.5mg/kg Q2W (PKAS) | Cohort I Efficacy Phase rHGG 4.5mg/kg Q2W (PKAS)
Number analyzed (Participants) | 3 | 5 | 3 | 5 | 9 | 4 | 12 | 7 | 6 | 1
mg/L
  Ctrough - after 1st dose: number analyzed (Participants) | 3 | 5 | 3 | 5 | 8 | 4 | 11 | 5 | 6 | 1
  Ctrough - after 1st dose | 16.7 [14.0 to 16.8] | 23.9 [21.1 to 27.2] | 33.8 [27.9 to 36.5] | 28.5 [19.6 to 42.2] | 48.3 [32.9 to 63.8] | 39.7 [33.9 to 41.9] | 26.0 [17.4 to 36.3] | 36.3 [25.2 to 178] | 35.8 [32.4 to 49.6] | NA [38.5 to 38.5] — n=1
  Ctrough - Week 16 (Cycle 4 Day 1) (4 weeks per cycle): number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 4 | 7 | 5 | 5 | 1
  Ctrough - Week 16 (Cycle 4 Day 1) (4 weeks per cycle) | NA [39.4 to 39.4] — n=1 | NA [78.6 to 78.6] — n=1 |  | NA [66.1 to 66.1] — n=1 | NA [66.1 to 66.1] — n=1 | 82.4 [65.7 to 104] | 94.3 [84.5 to 247] | 78.5 [57.0 to 134] | 122 [13.1 to 159] | NA [70.0 to 70.0] — n=1

13. Primary Outcome: Peak Concentration (Cmax) of Functional Cemiplimab (REGN2810) in Serum
Description: Cmax (peak concentration) of functional cemiplimab in serum reported.
Time Frame: Up to Week 16
Population: as for outcome 12
Measure: Median (Full Range); unit: mg/L
Arm/Group | Cohort A Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort B Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort D Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 4.5mg/kg Q2W (PKAS) | Cohort F Efficacy Phase ndDIPG 3mg/kg Q2W (PKAS) | Cohort H Efficacy Phase ndHGG 3mg/kg Q2W (PKAS) | Cohort J Efficacy Phase rHGG 3mg/kg Q2W (PKAS) | Cohort E Efficacy Phase ndDIPG 4.5mg/kg Q2W (PKAS) | Cohort I Efficacy Phase rHGG 4.5mg/kg Q2W (PKAS)
Number analyzed (Participants) | 3 | 5 | 3 | 5 | 9 | 4 | 12 | 7 | 6 | 1
mg/L
  Cmax - after 1st dose | 58.2 [52.0 to 86.9] | 73.5 [63.4 to 87.9] | 92.2 [87.9 to 101] | 68.3 [60.9 to 101] | 152 [76.0 to 202] | 95.1 [65.5 to 106] | 71.8 [6.41 to 88.0] | 88.8 [69.5 to 124] | 105 [93.7 to 130] | NA [123 to 123] — n=1
  Cmax -Week 16 (Cycle 4 Day 1) (4 weeks per cycle): number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 4 | 8 | 5 | 5 | 1
  Cmax -Week 16 (Cycle 4 Day 1) (4 weeks per cycle) | NA [122 to 122] — n=1 | NA [136 to 136] — n=1 | NA [112 to 112] — n=1 | NA [112 to 112] — n=1 | NA [236 to 236] — n=1 | 221 [164 to 256] | 165 [143 to 200] | 179 [119 to 234] | 209 [99.2 to 297] | NA [225 to 225] — n=1

14. Primary Outcome: Area Under the Concentration-time Curve (AUC) of Functional Cemiplimab (REGN2810) in Serum
Time Frame: Up to 24 months
Population: Cohorts used for pharmacokinetic endpoints were based on age and/or tumor type; Due to sparse sampling, area under the curve could not be calculated.
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Cohort A Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort B Phase 1 ST 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort D Phase 1 CNS 3mg/kg Q2W (PKAS) | Cohort C Phase 1 CNS 4.5mg/kg Q2W (PKAS) | Cohort F Efficacy Phase ndDIPG 3mg/kg Q2W (PKAS) | Cohort H Efficacy Phase ndHGG 3mg/kg Q2W (PKAS) | Cohort J Efficacy Phase rHGG 3mg/kg Q2W (PKAS) | Cohort E Efficacy Phase ndDIPG 4.5mg/kg Q2W (PKAS) | Cohort I Efficacy Phase rHGG 4.5mg/kg Q2W (PKAS)
Number analyzed (Participants) | 3 | 5 | 3 | 5 | 9 | 4 | 12 | 7 | 6 | 1
mg*hr/L | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated. | NA [NA to NA] — Due to sparse sampling, area under the curve could not be calculated.

15. Primary Outcome: Percentage of Progression-free Survival (PFS) at 12 Months for Participants With Newly Diagnosed HGG (ndHGG)
Description: PFS was defined as the time from randomization to the date of the first documented tumor progression, as determined per Response Assessment in Neuro-Oncology (RANO)/Immunotherapy Response Assessment in Neuro-Oncology (iRANO) criteria, or death due to any cause.
Time Frame: At 12 months
Population: Only participants with newly diagnosed HGG (ndHGG) were assessed for this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy
Number analyzed (Participants) | 12
Percentage of Participants | 22.2 [3.4 to 51.3]

16. Primary Outcome: Percentage of Overall Survival (OS) at 12 Months for Participants With ndDIPG and Recurrent HGG (rHGG)
Description: OS was defined as the time from randomization to the date of death due to any cause. A participant who had not died was censored at the last date that participant was documented to be alive. 95% CI is based on Kaplan-Meier method.
Time Frame: Up to 12 months
Population: Only participants with ndDIPG and recurrent HGG (rHGG) were assessed for this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 6 | 5 | 1 | 8
Percentage of Participants | 0.0 [NA to NA] — NA = Insufficient number of participants with events | 40.0 [5.2 to 75.3] | 0.0 [NA to NA] — NA = Insufficient number of participants with events | 35.7 [5.2 to 69.9]

17. Secondary Outcome: Objective Response Rate (ORR) for Participants Who Have a Confirmed Complete Response (CR) or Partial Response (PR)
Description: ORR was defined as the percentage of participants who have a confirmed complete response (CR) or partial response (PR), as determined per standard criteria between the date of first study treatment and the date of the first objectively documented progression or the date of receiving another anti-cancer systemic therapy, whichever came first. Clopper-Person exact confidence interval
Time Frame: Approximately 24 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Newly Diagnosed HGG (ndHGG) (Efficacy Phase): CNS TUMOR <12 yr REGN2810 4.5mg/kg Phase 1 (Cohort C2) CNS TUMOR <12 yr REGN2810 4.5mg/kg (Q2W)
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | Newly Diagnosed HGG (ndHGG) (Efficacy Phase) | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
Number analyzed (Participants) | 3 | 5 | 3 | 9 | 5 | 6 | 5 | 12 | 1 | 8
Percentage of Participants | 0 [0.0 to 70.8] | 0 [0.0 to 52.2] | 0 [0.0 to 70.8] | 0 [0.0 to 33.6] | 0 [0.0 to 52.2] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 8.3 [0.2 to 38.5] | 0 [0.0 to 97.5] | 0 [0.0 to 36.9]

18. Secondary Outcome: Number of Participants With Anti-REGN2810 Antibodies (ADA)
Description: ADA status classified as: Positive; Pre-existing (baseline [BL] sample positive & all post BL ADA titers reported as < 9-fold BL titer value); Negative (all samples negative); ADA positive: Treatment-boosted (positive result at BL with ≥1 post BL titer result ≥9-fold BL titer value); Treatment-emergent (TE) (negative result or missing result at BL with ≥1 positive post BL result); TE: Persistent (positive result detected in ≥2 consecutive post BL samples separated by ≥ a 12/16-week post BL period with no ADA-negative results in-between, regardless of any missing samples; Indeterminate (positive result in last collection, regardless of any missing samples); Transient (not persistent or indeterminate, regardless of any missing samples)
Time Frame: 1st follow-up visit, approximately 25 months
Population: ADA analysis set (AAS): all treated participants who received any amount of cemiplimab (SAF) & had ≥1 non-missing ADA result following first dose of cemiplimab (based on actual treatment received [as treated]).
  By design, the study arms were expected to be reflective of tumor type/diagnosis
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: 3mg/kg Q2W (AAS): Participants received REGN2810 3 milligrams/kilogram (mg/kg) once every 2 weeks (Q2W); anti-drug antibody analysis set (AAS)
- Phase 1: 4.5mg/kg Q2W (AAS): Participants received REGN2810 4.5mg/kg Q2W; AAS
- Efficacy Phase: 3mg/kg Q2W (AAS): Participants received REGN2810 3mg/kg Q2W + radiation therapy (CRT or HYRT); AAS
- Efficacy Phase: 4.5mg/kg Q2W (AAS): Participants received REGN2810 4.5mg/kg Q2W + radiation therapy (CRT or HYRT); AAS
Arm/Group | Phase 1: 3mg/kg Q2W (AAS) | Phase 1: 4.5mg/kg Q2W (AAS) | Efficacy Phase: 3mg/kg Q2W (AAS) | Efficacy Phase: 4.5mg/kg Q2W (AAS)
Number analyzed (Participants) | 16 | 5 | 19 | 7
Participants
  Negative | 16 | 5 | 17 | 6
  Pre-existing immunoreactivity | 0 | 0 | 1 | 0
  Treatment-emergent (TE) response | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 90 days after the last dose of study treatment (up to 36 months)
Groups:
- SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg: Phase 1 SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg (Q2W)
- CNS TUMOR <12 yr REGN2810 3mg/kg: Phase 1 CNS TUMOR <12 yr REGN2810 3mg/kg (Q2W)
- CNS TUMOR <12 yr REGN2810 4.5mg/kg: Phase 1 CNS TUMOR <12 yr REGN2810 4.5mg/kg (Q2W)
- CNS TUMOR 12 to <18 yr REGN2810 3mg/kg: Phase 1 CNS TUMOR 12 to <18 yr REGN2810 3mg/kg (Q2W)
- rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation: Efficacy Phase rHGG >= 12 yr REGN2810 3mg/kg (Q2W) + Re-Irradiation
Arm/Group | SOLID TUMOR < 12 yr REGN2810 3mg/kg | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 3mg/kg | CNS TUMOR <12 yr REGN2810 4.5mg/kg | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/5 | 2/3 | 8/9 | 3/5 | 6/6 | 4/5 | 7/12 | 1/1 | 5/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/3 | 3/9 | 0/5 | 3/6 | 3/5 | 7/12 | 0/1 | 5/8
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 2/3 | 8/9 | 4/5 | 6/6 | 5/5 | 12/12 | 1/1 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOLID TUMOR < 12 yr REGN2810 3mg/kg (N=3) | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg (N=5) | CNS TUMOR <12 yr REGN2810 3mg/kg (N=3) | CNS TUMOR <12 yr REGN2810 4.5mg/kg (N=9) | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg (N=5) | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy (N=6) | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy (N=5) | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy (N=12) | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation (N=1) | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation (N=8)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
IIIrd nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Family stress (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOLID TUMOR < 12 yr REGN2810 3mg/kg (N=3) | SOLID TUMOR 12 to <18 yr REGN2810 3mg/kg (N=5) | CNS TUMOR <12 yr REGN2810 3mg/kg (N=3) | CNS TUMOR <12 yr REGN2810 4.5mg/kg (N=9) | CNS TUMOR 12 to <18 yr REGN2810 3mg/kg (N=5) | ndDIPG <12 yr REGN2810 4.5mg/kg + Radiotherapy (N=6) | ndDIPG >=12 yr REGN2810 3mg/kg + Radiotherapy (N=5) | ndHGG >=12 yr REGN2810 3mg/kg + Radiotherapy (N=12) | rHGG <12 yr REGN2810 4.5mg/kg + Re-Irradiation (N=1) | rHGG >= 12 yr REGN2810 3mg/kg + Re-Irradiation (N=8)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 2 (3) | 2 (4) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (6) | 1 (2) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 3 (7) | 2 (3) | 6 (7) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 5 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 6 (10) | 0 (0) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 6 (8) | 1 (2) | 6 (8)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (4) | 1 (1) | 1 (2)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 3 (7) | 5 (10) | 0 (0) | 4 (4)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3)
Accessory nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Auditory nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmetria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IIIrd nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (7) | 1 (2) | 1 (3) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (4)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 1 (3) | 0 (0) | 3 (4) | 1 (2) | 2 (8) | 1 (1) | 3 (6)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (5)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (7) | 1 (1) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 8 (9) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pupillary reflex impaired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 2 (2)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Family stress (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As all efficacy cohorts for this study have now been closed due to the futility criteria, Regeneron as Sponsor in collaboration with PNOC made a decision to close the study to further enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03690869/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT03690869/SAP_001.pdf